CLINICAL TRIAL: NCT03396627
Title: Müller's Muscle as a New Proprioceptive Organ Evidence From Immunohistochemical Staining and Electron Microscopy to Verify That the Upper Eyelid Müller's Muscle Contains Proprioceptive Innervation for Reflexive Correction of Eyelid Position
Brief Title: Müller's Muscle as a New Proprioceptive Organ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Guy Ben-Simon, MD, Head, oculoplastic unit, Sheba Medical Center
Other Study IDs: 4384-17-SMC
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Eyelid Movement Disorders; Eyelid Ptosis Congenital
Keywords: eyelid; Muller

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — specimens of muller muscle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- muller muscle: muller muscle and conjunctiva excised during muller muscle conjunctival resection
  Interventions: Diagnostic Test: pathological examination

INTERVENTIONS:
Diagnostic Test: pathological examination — fresh MM specimens from patients undergoing Müllerectomies will undergo histologic examinations

SUMMARY:
Objectives: Upper eyelid retraction was believed to be maintained solely by voluntary contraction of the levator palpebrae superioris (LPS) and frontalis muscles, together with involuntary contraction of the sympathetically innervated Müller's muscle (MM). However, several studies have suggested that the LPS also undergoes involuntary contractions, and that a visual stimulus may not be the only trigger for frontalis muscle contractions. Recent studies hypothesized that the MM contains proprioceptive neuronal structures, which elicit involuntary LPS muscle contraction by the mesencephalic trigeminal nucleus via a continuous stretch reflex. We aim to identify proprioceptive structures in MM by means of histological examinations.

Methodology: Prospective study. Collaboration of oculoplastics, ophthalmologists and a neuroanatomy specialist in Sheba Medical Center. 50 fresh MM specimens from patients undergoing Müllerectomies will undergo histologic examinations, including immunohistochemical staining and light and electron microscopy.

Significance: Identification of proprioceptive structures in MM will be the first evidence-based proof of a proprioceptive mechanism in the eyelid. This might have a significant impact on future surgical management of eyelid procedures. Comprehensive understanding of the mechanisms underlying eyelid function is especially important in the management of children with ptosis who may have coexisting amblyopia.

DETAILED DESCRIPTION:
The investigators' goal is to find proprioceptive neuronal structures in Müller's muscle (MM). The investigatorswill recruit 50 MM specimens of patients diagnosed with either unilateral or bilateral ptosis who were referred to undergo a posterior approach surgical correction (MMCR). In this surgical approach, the proximal part of MM is removed between the levator palpebrae superioris muscle and the tarsus of the upper eyelids. The excised tissue is generally not used but simply discarded. For study purposed, the investigators will obtain the patients' consent to save these tissues and carry out histologic examinations of the samples. No change in the surgical procedure or the following management will be needed.

ELIGIBILITY:
Inclusion Criteria:

* specimens from patients undergoing Müllerectomies

Exclusion Criteria:

* small specimens (<1 cm length and width)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over 18 years old undergoing Müllerectomies
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2020-01-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
presence of proprioceptive organs in the muller muscle | 2 years
  presence of proprioceptive organs in the muller muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba_Medical_Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben Simon GJ, Blaydon SM, Schwarcz RM, Nakra T, Goldberg RA, McCann JD. Paradoxical use of frontalis muscle and the possible role of botulinum a toxin in permanent motor relearning. Ophthalmology. 2005 May;112(5):918-22. doi: 10.1016/j.ophtha.2005.01.004. PMID 15878076